CLINICAL TRIAL: NCT01475968
Title: Physiological Changes in Adults With Metabolic Syndrome Exposed to Concentrated Ultrafine Chapel Hill Air Particles
Brief Title: Physiological Changes in Adults With Metabolic Syndrome Exposed to Ultrafine Air Particles
Acronym: XCON
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: David Diaz-Sanchez (U.S. Federal Agency)
Collaborators: Environmental Protection Agency (EPA) (U.S. Federal Agency)
Responsible Party: Sponsor-Investigator, David Diaz-Sanchez, Biologist, Environmental Protection Agency (EPA)
Organization: Environmental Protection Agency (EPA) (U.S. Federal Agency)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: XCON; 04-1677 (Other: UNC IRB)
Record Dates: First submitted 2011-11-14; First posted 2011-11-22 (Estimated); Last update posted 2013-11-07 (Estimated); Status verified 2013-11

CONDITIONS: Metabolic Syndrome
MeSH Terms: conditions — Metabolic Syndrome | interventions — Particulate Matter; Environment, Controlled

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ultrafine Air Pollution Particulate Matter (Active Comparator): <2.5 microns concentrated from outside ambient air
  Interventions: Other: Ultrafine Air Pollution Particulate Matter
- Filtered Air (Sham Comparator): Filtered Air
  Interventions: Other: Filtered Air

INTERVENTIONS:
Other: Ultrafine Air Pollution Particulate Matter — Ultrafine (particle diameter less than 2.5 microns) Air Pollution Particulate Matter, concentrated from the ambient air outside of the Chapel Hill EPA Human Studies Facility
  Other Names: ultrafine particulate matter; concentrated ambient particulates (CAPS)
  Arms: Ultrafine Air Pollution Particulate Matter
Other: Filtered Air — Filtered Air
  Other Names: clean air
  Arms: Filtered Air

SUMMARY:
The purpose of this study is to examine the acute health effects of concentrated ambient ultrafine (UF) particulate matter (PM) exposure in patients with metabolic syndrome. Without lifestyle changes or medical intervention these patients are at considerable risk for developing diabetes and cardiovascular disease. Subjects (25-70) were exposed to both UF PM and filtered air for 2hr (at least 2 week interval), physiologic endpoints were measure pre-, post-, and 20hr post-exposure. Our hypothesis is that PM exposure in this population will result in changes in vascular and endothelial response as assessed by flow-mediated dilatation of the brachial artery and various heart rate variability and blood endpoints. This study and similar studies of susceptible populations are needed to provide the EPA with information regarding the health risks associated with ambient levels of UF PM.

ELIGIBILITY:
Inclusion Criteria:

* Age between 25-70 years old
* Metabolic syndrome as defined by the participant having at least three of the following criteria:

  * Abdominal obesity: Men waist circumference >102 cm (>40 in) Women waist circumference >88 cm (>35 in)
  * Triglycerides: ≥150 mg/dL
  * HDL cholesterol: Men <40 mg/dL and Women <50 mg/dL
  * Blood pressure: ≥130/≥85 mmHg OR have a history of high blood pressure requiring medication
  * Fasting glucose: ≥100 mg/dL and ≤126 mg/dL
* Normal resting electrocardiograph (ECG).

Exclusion Criteria:

* Current smoker or smoking history within 3 months of study (defined as more than one pack of cigarettes in the past 3 months).
* Oxygen saturation below 95% at the time of physical exam.
* Blood pressure ≥160/≥100 mmHg
* Fasting blood glucose >126 mg/dl
* Hypersensitivity to nitroglycerin or other nitrates
* Any chronic medical condition including active pulmonary disease, cardiovascular disease (coronary artery disease, heart failure, rhythm disturbances, etc.), neurological disease, liver disease, kidney disease, muscular disease, diabetes, other endocrine disease, hematologic/lymphatic disease, immune deficiency or autoimmune disease.
* Medications specifically prohibited include nitrates or other vasodilators (exception here includes erectile dysfunction medications if the participant agrees to refrain for 96 hours prior to study), anti-arrhythmics, physician prescribed anti-inflammatory agents, physician prescribed antioxidants, insulin and other medications for the treatment of diabetes. Participants must refrain from all over-the-counter anti-inflammatory agents, including aspirin, ibuprofen, and naproxen, and anti-oxidants for a period of one week prior to exposure. Low dose aspirin and statin regimens are acceptable. Medications not specifically mentioned here may be reviewed by the investigators prior to a participant's inclusion in the study. Additionally, medication regimens must remain constant during the study.
* Hepatitis B carriers
* Skin diseases or sensitivity precluding the use of ECG electrodes
* Active cancer, history of cancer within the last 5 years, untreated cancer. Potential participants may have a history of mild, treated skin cancer provided the condition does not interfere with ECG electrode placement.
* No exposure will be conducted within 4 weeks of a respiratory tract infection.
* History of serve migraines
* Pregnant women or nursing mothers

Ages: 25 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2004-12; Primary Completion 2011-06 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Changes in Vascular Function | change from baseline 0 hr after exposure, and change from baseline 20 hr after exposure. There will be at leat 2 weeks between the exposures
  1. Measurement of dilatation of the brachial artery (flow mediated and nitroglycerin mediated)
  2. Measurement of vasoconstrictor/vasodialtor, pro-coagulant, or pro-inflammatory mediators into systemic circulation (by ELISA of plasma)
  3. Measurement of changes in plasma levels of circulating microparticles and endothelial progenitor cells (as indicators of vascular injury or remodeling)

SECONDARY OUTCOMES:
Changes in heart rate variability | change from baseline 0 hr after exposure, and change from baseline 20 hr after exposure. There will be at leat 2 weeks between the exposures
  10 minute electrocardiogram recording (measure by Holter ECG) in which the subject has been resting for 20 minutes prior. Collected on a Mortara H12+ 12-Lead ECG Recorder (Mortara Instrument, Inc., Milwaukee, WI). The digitally recorded ECGs were sampled at 180 Hz and all data were stored on flash cards before processing.

CONTACTS AND LOCATIONS:
Overall Officials: Robert B Devlin, PhD, Principal Investigator — US EPA; Candice B Smith, PhD, Principal Investigator — US EPA
Locations (1):
- EPA Human Studies Facility, Chapel Hill, North Carolina, United States